CLINICAL TRIAL: NCT04029623
Title: Partnered Rhythmic Rehabilitation for Enhanced Motor-Cognition in Prodromal Alzheimer's Disease
Brief Title: Partnered Rhythmic Rehabilitation in Prodromal Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Madeleine Eve Hackney, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00110350; 1R01AG062691 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Prodromal Alzheimer's Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Partnered Rhythmic Rehabilitation (PRR) (Experimental): Participants in this study are will receive the PRR intervention. Participants will have two phases of intervention. In the three-month Training phase, participants will be assigned to 20, biweekly (90-minute) lessons over 12 weeks. In the nine-month Maintenance phase, participants will attend weekly lessons at least 3 times per month.
  Interventions: Other: Partnered Rhythmic Rehabilitation (PRR)
- Group walking (WALK) (Active Comparator): Participants in this study are will receive the WALK intervention. Participants will have two phases of intervention. In the three-month Training phase, participants will be assigned to 20, biweekly (90-minute) lessons over 12 weeks. In the nine-month Maintenance phase, participants will attend weekly lessons at least 3 times per month.
  Interventions: Other: Group walking (WALK)

INTERVENTIONS:
Other: Partnered Rhythmic Rehabilitation (PRR) — Partnered Rhythmic Rehabilitation (PRR) is moderate intensity, cognitively-engaging social dance that targets postural control systems. PRR involves learning complex stepping patterns and fosters tactile communication of motor goals between partners, enhancing social interaction's effect on cognition. Class sizes will consist of 10 or fewer pairs of participants with pAD and partners to maximize safety. Participants will engage in partnering exercises on how to interpret motor goals through touch, exercises to develop understanding of temporal relationship of movement to music, novel step introduction, connecting previously learned and novel step elements. Classes include practicing previously-learned steps, a 20-minute standing warm-up, and partnering and rhythmic enhancement exercises.
  Arms: Partnered Rhythmic Rehabilitation (PRR)
Other: Group walking (WALK) — WALK sessions consist of 10 minutes of warm-up, and evaluation/tips for practicing safe walking form mechanics (i.e., head up, shoulders relaxed, abdominals engaged, heel strike, roll and toe off; keep natural stride length, and speed up cadence if increased speed is desired), 55 minutes of walking with breaks, and 20 minutes of balance and stretching. WALK will take place in small groups with research assistants and trained family members and/or caregivers to control for social effects/contact of intervention. Participants of similar walking abilities will be 'buddied' with research assistants and trained physical therapy students who will act as group backmarkers, although participants will lead the pace. WALK participants will keep walking logs documenting their progress. WALK is expected to expend 3 metabolic equivalents (METs), like that of PRR.
  Arms: Group walking (WALK)

SUMMARY:
Interventions that affect many different aspects of human ability rather than just one aspect of human health are more likely to be successful in preventing and treating Alzheimer's disease (AD). Functional decline in AD is severely impacted by impaired ability to do physical actions while having to make decisions and concentrating, something scientists call motor-cognitive integration. Combined motor and cognitive training has been recommended for people with early AD, thus this study will use partnered, rhythmic rehabilitation (PRR), as an intervention to simultaneously target cardiovascular, social and motor-cognitive domains important to AD. PRR is moderate intensity, cognitively-engaging social dance that targets postural control systems, involves learning multiple, varied stepping and rhythmic patterns, and fosters tactile communication of motor goals between partners, enhancing social interaction's effect on cognition. Previous research demonstrates that PRR classes are safe and result in no injurious falls.

This study is a 12-month long Phase II single- blind randomized clinical trial using PRR in 66 patients with early AD. Participants with early AD will be randomly assigned to participate in PRR or a walking program for three months of biweekly sessions, followed by nine months of weekly sessions of PRR or walking. The overarching hypothesis is that PRR is safe, tolerable and associated with improved motor-cognitive function, and brain (neuronal), vascular (blood vessels) and inflammatory biomarkers that might affect function.

DETAILED DESCRIPTION:
For people with early Alzheimer's disease (AD), treatment options to prevent declined function are extremely limited, because AD affects many areas of function. In early AD, people may have trouble physically doing things while also thinking, which is necessary for many activities in daily life. This problem might be helped by doing activities that challenge the mind and the body at the same time. Partnered rhythmic rehabilitation (PRR), which targets fitness, cognition, mobility and social engagement and may prevent future functional problems in AD.

This is a phase II single-blind randomized clinical trial to assess the safety, tolerability, and efficacy of PRR in individuals in the early stages of AD, also called prodromal AD (pAD) . Participants will be randomly assigned to 90-minute PRR or WALK classes. Both interventions will receive equal contact and monitoring from study staff. Participants will have two phases of intervention. In the three-month Training phase, participants will be assigned to 20, biweekly (90-minute) lessons over 12 weeks. In the nine-month Maintenance phase, participants will attend weekly lessons at least 3 times per month. Participants will undergo either PRR or Walking Exercise (WALK) interventions for one year, which will use de-escalating doses: two times per week for three months (Training) and weekly for nine months (Maintenance).

The first study aim is to determine acceptability, safety, tolerability and satisfaction with PRR in pAD. The second aim is to determine a) efficacy of PRR vs. WALK for improving motor-cognitive integration in pAD; b) to identify sensitive endpoints to power a future phase III trial. The researchers will also explore potential mechanisms by which PRR affects pAD. These mechanisms include functional brain measures, vascular, and inflammation measures (arterial stiffness; cerebral perfusion, task functional magnetic resonance imaging [fMRI]; inflammatory markers: cytokines and chemokines, endothelial adhesion markers.

ELIGIBILITY:
Inclusion Criteria:

* Amnestic mild cognitive impairment (MCI) will be defined using the AD Neuroimaging Initiative (ADNI) criteria (http://www.adni-info.org/Scientists/ADNIStudyProcedures.aspx). All MCI participants in ADNI are required to have an amnestic subtype defined as:

  * Subjective memory concern or a memory problem noted by their partner
  * Abnormal memory function documented by a specified education adjusted cutoff score on the delayed paragraph recall of the Anna Thompson story of the Logical Memory subtest from the Wechsler Memory Scale-Revised
  * Mini-Mental State Exam (MMSE) score between 24 and 30 (inclusive). Exceptions may be made for subjects with less than 8 years of education at the discretion of the PI
  * Single or multi-domain amnestic MCI (both subtypes are at high risk for progression to AD)
  * Clinical Dementia Rating (CDR) = 0.5 (Memory Box score must be at least 0.5)
  * General functional performance sufficiently preserved
* Ability to walk 10 or more feet without an assistive device
* Completed six grades of education or has a good work history (sufficient to exclude intellectual disabilities)
* Achieves less than 150 minutes of moderate intensity or 75 minutes of vigorous intensity aerobic activity per week, which is the recommended amount of weekly exercise as per the US Department of Health and Human Services. Not involved in any structured exercise program within the past 3 months (brisk walks are considered formal exercise but leisurely walks are not)
* Not hospitalized within the last 60 days
* Willing to commit to a one year research program

Exclusion Criteria:

* Acute medical illness requiring hospitalization
* Uncontrolled congestive heart failure
* History of stroke in the past three years
* Inability to perform study procedures
* Inability to perform MRI (e.g. metal implants or cardiac pacemaker, claustrophobia)
* Medical or physical conditions that would preclude participation (e.g., severe arthritis or mobility problems, uncontrolled hypertension or diabetes, renal failure, history of angina with activity)
* On medications that could adversely affect cognition, eg: antipsychotics, opioids, stimulants, chemotherapy, anti-parkinsonian drugs (eg Levodopa), neurologic prescriptions to treat Multiple sclerosis and/or Parkinson's. Patients will also be excluded if they are not on stable doses of Aricept, or anticholinesterase inhibitors, eg Namenda, for at least 3 months
* Psychotic disorders
* Confounding neurologic conditions (e.g., active central nervous system (CNS) opportunistic infections, seizure disorders, head injury with loss of consciousness >30 minutes, intracranial neoplasms, stroke with neurological or neuropsychiatric sequelae)
* Substance Use Disorder, Major Depressive and Generalized Anxiety Disorders within six months of evaluation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Four Square Step Test (FSST) Time | Baseline, 3 months, 12 months
  The Four Square Step Test (FSST) assesses mechanisms underlying motor-cognitive integration. FSST requires participants to step clockwise then counterclockwise into four squares created by rods arranged on the ground in a cross. Participants are instructed to perform FSST "as quickly and as safely as you can," to not touch the rods and make both feet contact the floor in each square. Timing begins when the participant initiates movement and stops when both feet are back in the starting square after completing the sequence. Trials will be repeated if the participant does not understand the instructions, fails to complete the sequence accurately, loses balance, or touches a rod. Three successful trials will be recorded and fastest time selected for analyses.
Change in Acceptability | Baseline, Month 12
  Acceptability of the intervention will be assessed by conducting two pre-session focus groups with 8-10 pAD participants. Focus groups will assess barriers and facilitators of PRR as therapy for motor-cognitive performance of functional activity issues. Post training, the researchers will conduct two focus groups with 8 participants each to assess satisfaction with PRR, perceived effect of PRR on participation in life's activities, impact of touch on therapy, overall perceived impact of cognitive impairment on benefits/results from PRR, and solicit recommendations for improvement. Responses will be open ended rather than on a pre-determined scale.
Number of Injurious Falls | Month 12
  The primary safety outcome is the number of injurious falls as a result of participation in PRR. PRR will be considered safe if no injurious falls are observed during PRR instruction.
Attrition | Month 12
  Tolerability will be assessed by the number of participants completing the study. PRR will be considered tolerable if attrition is less than or equal to 15 percent.

SECONDARY OUTCOMES:
Change in Timed Up and Go (TUG) Test - Cognitive Time | Baseline, 3 months, 12 months
  For the TUG-Cognitive test, participants must pay attention to walking and counting. Participants are instructed to stand up from a chair, walk 3 meters as quickly and safely as possible, cross a line marked on the floor, turn around, walk back, and sit down; at the same time they are asked to count backward by threes from a randomly selected number between 20 and 100. Participants are timed (in seconds) beginning when the test administrator says "go" and ending when the participant completed the task and sits down.
Change in Body Position Spatial Task (BPST) | Baseline, 3 months, 12 months
  Body Position Spatial Task (BPST), is a validated visuospatial memory task. The BPST incorporates spatial memory and navigational skills while maintaining posture. The examiner verbally and visually shows a series of side, forward and turning steps, which the examinee repeats. If the examinee repeats the entire pattern correctly they are scored with a 1; any incorrect parts of the pattern mean the score will be 0. Participants complete up to 8 different sequences, and have up to 2 tries to perform the sequence correctly. Total scores can range from 0 to 8, with higher values indicating more sequences correctly performed.
Change in Lawton Instrumental Activities of Daily Living (IADL) Score | Baseline, 3 months, 12 months
  Functional independence will be measured with the Instrumental Activities of Daily Living (IADL) scale. The IADL is an 8-item instrument which assesses how well the respondent can perform daily tasks by rating the responses as 0 or 1. The total score ranges from 0 to 8, with higher scores indicating greater independence.
Change in Composite Physical Function (CPF) Scale Score | Baseline, 3 months, 12 months
  Functional independence will be measured with the Composite Physical Function (CPF) Scale. The CPF has 12 items where respondents rate how well they can perform certain tasks on a scale of 0 (cannot do) to 2 (can do on own without help). Total scores range from 0 to 24, with higher scores indicating better ability to perform activities without assistance.
Change in Short Physical Performance Battery (SPPB) Score | Baseline, 3 months, 12 months
  The SPPB asks participants to perform movements to assess balance, gait, and lower extremity strength and endurance. Total scores range from 0 to 12, with higher scores indicating better physical performance.
Change in Mini-Balance Evaluation Systems Test (Mini-BESTest) Score | Baseline, 3 months, 12 months
  This clinical balance assessment tool is a shortened version of the Balance Evaluation Systems Test (BESTest). It aims to target and identify 6 different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits. The Mini-BESTest has 14 items that are scores on a scale of 0 (lowest level of function) to 2 (highest level of function). Total scores range from 0 to 28 where higher scores indicate better function.
Change in 6 Minute Walk Test (6MWT) Distance | Baseline, 3 months, 12 months
  The 6 minute walk test (6MWT) assesses distance, in meters, walked over 6 minutes as a sub-maximal test of aerobic capacity and endurance.
Change in Preferred Gait Speed | Baseline, 3 months, 12 months
  Gait speed testing will be administered using a GAITRite walkway. GAITRite is a pressure sensitive walkway that can assess gait anomalies. Gait speed while participants walk at their preferred speed will be compared between study arms.
Change in Backward Gait Speed | Baseline, 3 months, 12 months
  Gait speed testing will be administered using a GAITRite walkway. GAITRite is a pressure sensitive walkway that can assess gait anomalies. Gait speed while walking backwards will be compared between study arms.
Change in Fast Gait Speed | Baseline, 3 months, 12 months
  Gait speed testing will be administered using a GAITRite walkway. GAITRite is a pressure sensitive walkway that can assess gait anomalies. Gait speed while walking as fast as possible will be compared between study arms.
Change in Clinical Dementia Rating (CDR) Questionnaire Score | Baseline, 3 months, 12 months
  The CDR is designed to reflect level of cognitive impairment based on a semi-structured interview with an informant and a separate mental status exam with the patient. The clinician rates each of the six general domains involving memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care. A global rating is then generated, ranging from 0-no impairment to 3-severe impairment.
Change in Flanker Task Score | Baseline, 3 months, 12 months
  The Flanker Task of the Executive Abilities Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER) instrument involves responding to a central stimulus while ignoring flanking stimuli that are either compatible or incompatible with the central stimulus. Composite scores range from 1 to 10, where higher scores indicate faster and more accurate reactions.
  The EXAMINER is a 30-40 minute test battery funded with support from the NIH that reliably and validly assesses executive function in clinical trials. This computer administered instrument assesses working memory, response inhibition, set shifting, and phonemic and category fluency.
Change in Set Shifting Score | Baseline, 3 months, 12 months
  The Set Shifting assessment of the EXAMINER instrument is a measure of mental flexibility assessing the subject's ability to attend to the specific attributes of compound stimuli, and to shift that attention when required. Participants match shapes or colors, as instructed, and composite scores range from 1 to 10, where higher scores indicate greater accuracy.
  The EXAMINER is a 30-40 minute test battery funded with support from the NIH that reliably and validly assesses executive function in clinical trials. This computer administered instrument assesses working memory, response inhibition, set shifting, and phonemic and category fluency.
Change in Spatial 1-Back Test Score | Baseline, 3 months, 12 months
  The Spatial 1-Back Test of the EXAMINER instrument assesses spatial working memory. The spatial 1-back test has 30 trials where the number of correct "yes" or "no" responses are tabulated. The total number of correct responses ranges from 0 to 30 with higher scores indicating greater accuracy.
  The EXAMINER is a 30-40 minute test battery funded with support from the NIH that reliably and validly assesses executive function in clinical trials. This computer administered instrument assesses working memory, response inhibition, set shifting, and phonemic and category fluency.
Change in Dot Counting Test Score | Baseline, 3 months, 12 months
  The Dot Counting Test of the EXAMINER instrument assesses verbal working memory. The dot counting test includes 6 trials, which progress in difficulty, where participants count dots. Scoring is based on the participant's ability to correctly recall the number of dots they counted. The total number of correct responses ranges from 0 to 27 with higher scores indicating greater accuracy in recall.
  The EXAMINER is a 30-40 minute test battery funded with support from the NIH that reliably and validly assesses executive function in clinical trials. This computer administered instrument assesses working memory, response inhibition, set shifting, and phonemic and category fluency.
Change in Verbal Fluency Test Score | Baseline, 3 months, 12 months
  The Verbal Fluency Test of the EXAMINER instrument uses list generation which requires participants to generate words beginning with a specific letter, and category fluency in which the participant generates words from a specified category (e.g., animals, fruits). There are four 1-minute trials where participants name as many items as they can (up to 40) that fit the requested criteria. Total scores range from 0 to 160, where higher values mean that more words fitting the criteria provided.
  The EXAMINER is a 30-40 minute test battery funded with support from the NIH that reliably and validly assesses executive function in clinical trials. This computer administered instrument assesses working memory, response inhibition, set shifting, and phonemic and category fluency.
Change in Reverse Corsi Blocks Levels Completed | Baseline, 3 months, 12 months
  Spatial cognition will be assessed by administration of the Reverse Corsi Blocks in which the examiner taps a series of blocks and the participant then produces this pattern but in the opposite order. Up to eight different levels, with increasingly difficult patterns, are performed. The total score for the exam ranges from 1 to 9, with higher values indicating more levels successfully performed.
Change in Patient Health Questionnaire (PHQ-9) Score | Baseline, 3 months, 12 months
  The Patient Health Questionnaire (PHQ-9) is a 9-item, validated measure of depression severity in dementia. Respondents indicate how bothered by problems they are on a scale from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 27, where higher scores indicate more severe depression.
Change in Multidimensional Scale of Perceived Social Support (MSPSS) Score | Baseline, 3 months, 12 months
  The MSPSS has 12 items assessing how social support factors are perceived by individuals. This scale has three subscales to evaluate support by family, friends and significant others. Respondents rate statements on a scale of 1 (very strongly disagree) to 7 (very strongly agree). Total scores range from 12 to 84, where higher scores indicate increased perception of social support.
Change in Montreal Cognitive Assessment (MoCA) Score | Baseline, 3 months, 12 months
  MoCA is an instrument to screen for mild cognitive dysfunction, assessing the cognitive domains of attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Total scores range from 0 to 30 with higher scores indicating better cognitive function. A normal score is considered to be 26 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Hackney, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available for sharing after deidentification.
Time Frame: Data will be shared one year after study publication.
Access Criteria: Researchers requesting individual participant data will be asked to sign a data use agreement prior to accessing the data. Data can be requested by contacting Dr. Hackney at mehackn@emory.edu